CLINICAL TRIAL: NCT02598622
Title: A Phase II Pilot Study Investigating the Effects of Acetyl-L-Carnitine and Vincristine-Induced Neuropathy in Pediatric Patients With ALL
Brief Title: A Pilot Study Investigating the Effects of Acetyl-L-Carnitine and Vincristine-Induced Neuropathy in Pediatric Patients With ALL
Acronym: ALC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug availability
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Chie-Schin Shih, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1011003177
Record Dates: First submitted 2015-08-25; First posted 2015-11-06 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Vincristine Induced Neuropathy
MeSH Terms: interventions — Acetylcarnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetyl-L-Carnitine only (Experimental): The first 15 subjects participating in this study will receive Acetyl-L-Carnitine and pharmacokinetic testing will be done.
  Interventions: Drug: Acetylcarnitine
- Acetyl-L-Carnitine or Placebo (Experimental): Subjects 16-30 will be randomized to receive drug or placebo.
  Interventions: Drug: Acetylcarnitine; Drug: Placebo

INTERVENTIONS:
Drug: Acetylcarnitine — Acetylcarnitine is taken 2 times a day for days 1 through 21.
Drug: Placebo — Placebo is taken 2 times a day for days 1 through 21.
  Arms: Acetyl-L-Carnitine or Placebo

SUMMARY:
The purpose of this study is to see if a drug called Acetyl-L-Carnitine can help prevent painful nerve damage and nerve pain which is caused by vincristine, a drug used in chemotherapy in children being treated for newly diagnosed ALL. Acetyl-L-Carnitine is a drug available for purchase as a nutritional supplement but for the purpose of this study is experimental.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following inclusion criteria.

  * The subject must have a confirmed diagnosis of acute lymphoblastic leukemia within 1 week of starting therapy
  * Currently being treated on a standard ALL induction regimen
  * Subjects must be greater than or equal to 5 and less than 18 years old
  * Signed informed consent

Exclusion Criteria:

* Subjects will be excluded for the following:

  * Preexisting neurologic disease, including grade II, III, or IV neurological status by NCI Common Toxicity Criteria v3.0 on clinical exam
  * History of hypersensitivity to vincristine
  * History of hypersensitivity to Acetyl-L-carnitine
  * Previous use of Acetyl-L-carnitine
  * Concurrent anti-convulsant use
  * Concurrent Gabapentin use
  * Concurrent Glutamine use
  * Liver Function: Total bilirubin greater than 1.3 mg/dL and serum glutamic-pyruvic transaminase (SGPT) (ALT) greater than 5 x upper limit of normal for age and serum albumin less than 2 g/dL
  * Patients who are pregnant

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2016-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetyl-L-Carnitine Only | Acetyl-L-Carnitine or Placebo
Started | 8 | 0 (Study terminated prior to randomization phase. No enrollment in this arm.)
Completed | 2 | 0
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetyl-L-Carnitine Only | Acetyl-L-Carnitine or Placebo | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 |  | 8
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Full Range); unit: years] | 8 [5 to 14] |  | 8 [5 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 |  | 5
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 |  | 3
  Not Hispanic or Latino | 5 |  | 5
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 8 |  | 8
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Grade of Neurotoxicity Will be Captured by an Adaptation of the Total Peripheral Neuropathy Score.
Time Frame: Days 1 - 21
Population: Only 2 out of 8 participants were able to complete protocol related therapy and therefore no data were collected for analysis.
Arm/Group | Acetyl-L-Carnitine Only | Acetyl-L-Carnitine or Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Acetyl-L-Carnitine Only | Acetyl-L-Carnitine or Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetyl-L-Carnitine Only (N=8) | Acetyl-L-Carnitine or Placebo (N=0)
Hospitalization (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetyl-L-Carnitine Only (N=8) | Acetyl-L-Carnitine or Placebo (N=0)
Low Hemoglobin (Blood and lymphatic system disorders) | 8 (16) | 0 (0)
Low Platelets (Blood and lymphatic system disorders) | 8 (14) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — short of breath
pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — hip pain
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — RASH ON HAND
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Unable to meet enrollment goals. Drug expired prior to being able to enroll total subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes